CLINICAL TRIAL: NCT04644484
Title: A Phase III Randomized Blinded Study to Evaluate SYN023 Compared to Human Rabies Immune Globulin in Post Exposure Prophylaxis of Rabies in Adults With Category III Rabies Exposure Risks
Brief Title: A Phase III Clinical Study to Evaluate SYN023's Efficacy and Safety
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Synermore Biologics (Suzhou) Co., Ltd. (Industry)
Collaborators: Simoon Record Pharma Information Consulting Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SYN023-006
Record Dates: First submitted 2020-11-16; First posted 2020-11-25 (Actual); Results first posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-03

CONDITIONS: Rabies; Communicable Disease; Virus Diseases; Rhabdoviridae Infections; Mononegavirales Infections; RNA Virus Infections
Keywords: Post-exposure prophylaxis of Rabies
MeSH Terms: conditions — Rabies; Communicable Diseases; Virus Diseases; Rhabdoviridae Infections; Mononegavirales Infections; RNA Virus Infections | interventions — Rabies Vaccines

STUDY DESIGN:
Intervention Model Description: In this study, 1000 subjects aged 18 and over who had Grade 3 exposure to rabies virus were intended to be enrolled, and randomly assigned to the experimental group and the control group (3:1). Both groups were immunized according to PEP procedures for rabies.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding for drugs were carried out by the randomization statistician and other personnel who will not be involved in the implementation of the clinical trial. Under the guidance of the randomization statistician, blinding operators attach the printed labels with numbers to the outer packages of the study drug/control drug according to the blind codes and seal the packages with sealing stickers.
  After the completion of blinding for drugs, the blind codes shall be sealed and kept by the randomization statistician. The entire blinding process must be documented. The personnel responsible for blinding must not participate in other relevant works during this clinical trial, and must not disclose the blind codes to any person participating in this clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Group: SYN023+Rabies Vaccine (Experimental): SYN023:
  Interventions: are administered by direct injection into the wound or by subcutaneous or intramuscular injection when this is not possible SYN023 is an equal mass mixture of CTB011 and CTB012, two monoclonal antibodies that exhibit a wide spectrum of activity against various wild-type rabies strains in vitro.
  Dosage form: 6mg/2mL, liquid; Dosage: 0.3 mg/kg of SYN023; Frequency/duration: at Day 1
  Rabies vaccine :
  Interventions: should be administered in deltoid muscle Dosage form: >=2.5 IU, freeze-dried vaccine, reconstitute into 0.5 mL before use Dosage: 0.5 mL after reconstitution Frequency/duration: at Day 1, 4, 8, 15, 29
  Interventions: Biological: SYN023; Biological: Rabies Vaccine
- Control Group: Human Rabies Immune Globulin (HRIG)+Rabies Vaccine (Active Comparator): Human Rabies Immune Globulin (HRIG):
  Interventions: are administered by direct injection into the wound or by subcutaneous or intramuscular injection when this is not possible Dosage form: 100 IU/mL, liquid; Dosage: 20 IU/kg; Frequency/duration: at Day 1
  Rabies vaccine :
  Interventions: should be administered in deltoid muscle Dosage form: >=2.5 IU, freeze-dried vaccine, reconstitute into 0.5 mL before use; Dosage: 0.5 milliliters (mL) after reconstitution; Frequency/duration: at Day 1, 4, 8, 15, 29
  Interventions: Biological: Human Rabies Immune Globulin (HRIG); Biological: Rabies Vaccine

INTERVENTIONS:
Biological: SYN023 — The finished product of SYN023 is a mixture of 3.0 mg/mL CTB011 and 3.0 mg/mL CTB012 at a ratio of 1:1. SYN023 is a sterile and preservative-free injection, and the excipient contains 25 mM histidine (3.879 mg/mL), 150 mM sodium chloride (8.766 mg/mL) and 0.02% polysorbate 80 (0.2 mg/mL) and pH of 6.0. Each vial contains 2.15 mL of SYN023, or 6.45 mg of monoclonal antibody. The glass bottle was closed with a 13 mm bromobutyl rubber stopper, a 13 mm aluminum crimping cap and a polypropylene flip-open lid.
  Other Names: A Humanized Anti-Rabies Molecular antibodies cocktails
  Arms: Experimental Group: SYN023+Rabies Vaccine
Biological: Human Rabies Immune Globulin (HRIG) — The HRIG is a Chinese licensed Human Rabies Immunoglobulin, which are derived from human plasma, and then purified and filled in the injectable vial form. The HRIG is indicated for the Post-exposure Prophylactic (PEP) of Rabies
  Arms: Control Group: Human Rabies Immune Globulin (HRIG)+Rabies Vaccine
Biological: Rabies Vaccine — Interventions: The Chinese licensed rabies vaccine should be administered in deltoid muscle Dosage form: >=2.5 IU, freeze-dried vaccine, reconstitute into 0.5 milliliters (mL) before use Dosage: 0.5 mL after reconstitution Frequency/duration: at Day 1, 4, 8, 15, 29
  Other Names: Freeze-dried Rabies Vaccine for Human Use (Vero Cells)

SUMMARY:
This is a Phase 3, blinded, randomized study of SYN023 compared to a China licensed Human Rabies Immunoglobulin (a Rabies immune globulin from human sources, HRIG) for the prevention of rabies as part of post-exposure prophylaxis (PEP). The trial will enroll the World Health Organization (WHO) Category III rabies exposure subjects. The subject's death and rabies data will be reviewed by Data and safety monitoring board (DSMB) to confirm the safety. Besides, rabies vaccine would be administered after Study Drug in each group.

This trial is proposed to further the licensure of SYN023 to provide an effective PEP alternative available to those exposed persons who need such a product. A placebo-controlled rabies trial is unethical thus HRIG is selected as the control group. Rabies immune globulin from equine and human sources (HRIG) have been evaluated in many trials and HRIG is the standard of care in China.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, blinded, and active controlled study of SYN023 compared with a China licensed HRIG for PEP of patients who have been confirmed to have met all inclusion/exclusion criteria for their treatment group.

1000 patients aged 18 and above with the World Health Organization (WHO) Category III rabies exposure should be enrolled as planned and randomly assigned to the experimental group and the control group based on a ratio of 3: 1 through on-site stratification as part of PEP.

All subjects should receive wound infiltration injection of SYN023 or HRIG on Study Day 1 (wound conditions should be described and recorded before injection, including diameter, depth, expansion treatment, etc.), and should also simultaneously receive intramuscular injection of one dose of the freeze-dried rabies vaccine for human use (Vero cells) into the deltoid muscle. In accordance with the Essen Scheme, each subject also needs to receive one dose of the freeze-dried rabies vaccine for human use (Vero cells) on Study Days 4, 8, 15, and 29 respectively.

3.0 mL of venous blood samples should be collected 8 times from each subject prior to administration and on Study Day 4, 8, 15, 43, 99, 183, and 365 post administration of study drug. Relevant information should be collected from the subjects through follow-up visits, such as occurrence of rabies and survival conditions.

RVNA should be assayed through rapid fluorescence focus inhibition test (RFFIT).

Local adverse events related to the SYN023 injection sites and injection sites of the first dose and second dose of rabies vaccine, and systemic adverse events (AE) other than injection sites should be collected within 7 days after administration; local adverse events related to the injection sites of the third dose, fourth dose and fifth dose of rabies vaccine, and systemic adverse events (AE) other than the injection sites should be collected 7 days after administration. In addition, all adverse events occurring within 43 days after administration should be collected, and pregnancy conditions in 6 months after administration and all serious adverse events (SAE) occurring during the study period should be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Is age ≥18 years, on Study Day 1 with legal identification documents, and plan to live in the local administration area during the study;
2. Category III rabies exposure within 24 hours before Study Drug receipt ;
3. Completed written informed consent process, and signed the informed consent forms;
4. Subjects with the ability to understand the study procedure. And agreed to complete all follow-ups;
5. Female subjects are not in pregnancy (with negative results of urine pregnancy tests before vaccination) and are not in the period of breast feeding, and agree to avoid pregnancy within 121 days after administration;
6. Those who have an armpit temperature ≤ 37.0 °C.

Exclusion Criteria:

1. Previous receipt of equine or human (rabies) globulin or rabies vaccination prior to randomization;
2. Clinical evidence of rabies infection;
3. Category I and Category II rabies exposure;
4. Had fever (armpit temperature ≥ 38.5 °C) within 3 days before Study Day 1, or in the acute episode of any chronic diseases;
5. Received immunoglobulin or blood products (except for the anti-tetanus immunoglobulin) within 43 days before Study Day 1, or plan to use any such product (except for the anti-tetanus immunoglobulin) during the study;
6. Received systemic immunosuppressant medication such as systemic corticosteroids but not limited to systemic corticosteroids within 43 days before Study Day 1;
7. History of any immunodeficiency disease (for example: AIDS, systemic lupus erythematosus, etc.); or Laboratory evidence of previous or current immunodeficiency disease, including, but not limited to, any laboratory evidence of HIV infection;
8. History of spleen function deficiency or function injury, such as no spleen caused by any cause (such as splenectomy);
9. History of any severe allergy for vaccination, such as systemic urticaria, allergic laryngeal edema, anaphylactoid purpura, local allergic necrosis (Arthus reaction), angioedema, anaphylactic shock, etc., or allergic to any ingredient of the study drug/vaccine;
10. Previous receipt of any study product (drug, vaccine, biological product or medical device) within 6 months before Study Day 1, or plan to participate in any other clinical study during this study period;
11. History of or clinical evidence of any systemic disease, acute disease or chronic disease (such as convulsions, epilepsy, encephalopathy, nephrotic syndrome, etc.) that the investigator considers to be likely to interfere with safety or efficacy assessment of the study;
12. Previous medical history that may compromise the safety of the subject in the study according to the opinion of the principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoqiang Liu, MD, PhD, Principal Investigator — Yunnan Province CDC
Locations (1):
- Yunnan Province Center for Disease Control and Prevention (CDC), Kunming, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McClain JB, Chuang A, Reid C, Moore SM, Tsao E. Rabies virus neutralizing activity, pharmacokinetics, and safety of the monoclonal antibody mixture SYN023 in combination with rabies vaccination: Results of a phase 2, randomized, blinded, controlled trial. Vaccine. 2021 Sep 24;39(40):5822-5830. doi: 10.1016/j.vaccine.2021.08.066. Epub 2021 Sep 3. PMID 34483020
- [Result] Ding Y, Wu M, Zhang H, Zhu X, Hu Y, Li X, Liu J, Tsao E, Liu M, Li C. Safety, pharmacokinetics and pharmacodynamics of SYN023 alone or in combination with a rabies vaccine: An open, parallel, single dose, phase 1 bridging study in healthy Chinese subjects. Antiviral Res. 2020 Dec;184:104956. doi: 10.1016/j.antiviral.2020.104956. Epub 2020 Oct 19. PMID 33091433
- [Derived] Liu X, Zha Y, Wang Z, Jiang Y, Zhang X, Guo J, Li J, Zhang Q, Tsao E. The pharmacokinetics and safety comparison of Zamerovimab and Mazorelvimab monoclonal antibodies vs. HRIG in category III rabies post-exposure prophylaxis: a stratified analysis by wound characteristics. Biologicals. 2025 Nov;92:101852. doi: 10.1016/j.biologicals.2025.101852. Epub 2025 Aug 13. PMID 40812204
- [Derived] Liu X, Li J, Zha Y, Wang Z, Jiang Y, Zhang X, Guo J, Yu J, Li X, Zhang Q, Reid C, McClain JB, Tsao E. The efficacy and safety of SYN023 (Zamerovimab and Mazorelvimab injection), the recombinant humanized anti-rabies virus monoclonal antibody mixture, combined with rabies vaccine in a WHO category III rabies post-exposure population: A randomized, double-blind, positive control, phase III clinical trial. Vaccine. 2025 Aug 13;61:127289. doi: 10.1016/j.vaccine.2025.127289. Epub 2025 Jun 5. PMID 40479926

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Group: SYN023+Rabies Vaccine: 1000 patients aged 18 and above with World Health Organization (WHO) Category III rabies exposure should be enrolled as planned and randomly assigned to the experimental group and the control group based on a ratio of 3:1 through on-site stratification as part of post-exposure prophylaxis (PEP).
  SYN023: 0.3 mg/kg, wound infiltration injection. If the study drug isn't used up after infiltration injection for all wounds, the remaining amount should be injected into the muscles far away from the vaccine injection sites Frequency/duration: at Day 1
  Rabies Vaccine: 0.5 milliliters (mL), intramuscular injection into the deltoid muscle Frequency/duration: at Day 1, 4, 8, 15, 29
- Control Group: Human Rabies Immune Globulin (HRIG)+Rabie Vaccine: 1000 patients aged 18 and above with World Health Organization (WHO) Category III rabies exposure should be enrolled as planned and randomly assigned to the experimental group and the control group based on a ratio of 3:1 through on-site stratification as part of post-exposure prophylaxis (PEP).
  Human Rabies Immune Globulin (HRIG): 20 IU/kg, wound infiltration injection. If the study drug isn't used up after infiltration injection for all wounds, the remaining amount should be injected into the muscles far away from the vaccine injection sites Frequency/duration: at Day 1
  Rabies Vaccine: 0.5 milliliters (mL), intramuscular injection into the deltoid muscle Frequency/duration: at Day 1, 4, 8, 15, 29
Period: Overall Study
Arm/Group | Experimental Group: SYN023+Rabies Vaccine | Control Group: Human Rabies Immune Globulin (HRIG)+Rabie Vaccine
Started | 750 | 250
Completed | 750 | 250
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental Group: SYN023+Rabies Vaccine: 1000 patients aged 18 and above with WHO Category III rabies exposure should be enrolled as planned and randomly assigned to the experimental group and the control group based on a ratio of 3:1 through on-site stratification as part of post-exposure prophylaxis (PEP).
  SYN023: 0.3 mg/kg, wound infiltration injection. If the study drug isn't used up after infiltration injection for all wounds, the remaining amount should be injected into the muscles far away from the vaccine injection sites Frequency/duration: at Day 1
  Rabies Vaccine: 0.5 milliliters (mL), intramuscular injection into the deltoid muscle Frequency/duration: at Day 1, 4, 8, 15, 29
- Control Group: Human Rabies Immune Globulin (HRIG)+Rabie Vaccine: 1000 patients aged 18 and above with WHO Category III rabies exposure should be enrolled as planned and randomly assigned to the experimental group and the control group based on a ratio of 3:1 through on-site stratification as part of post-exposure prophylaxis (PEP).
  Human Rabies Immune Globulin (HRIG): 20 IU/kg, wound infiltration injection. If the study drug isn't used up after infiltration injection for all wounds, the remaining amount should be injected into the muscles far away from the vaccine injection sites Frequency/duration: at Day 1
  Rabies Vaccine: 0.5 milliliters (mL), intramuscular injection into the deltoid muscle Frequency/duration: at Day 1, 4, 8, 15, 29
- Total: Total of all reporting groups
Arm/Group | Experimental Group: SYN023+Rabies Vaccine | Control Group: Human Rabies Immune Globulin (HRIG)+Rabie Vaccine | Total
Number analyzed (Participants) | 750 | 250 | 1000
Age, Continuous [Mean (Full Range); unit: years] | 43.7 [18 to 79] | 44.6 [19 to 86] | 43.9 [18 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 346 | 117 | 463
  Male | 404 | 133 | 537
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 750 | 250 | 1000
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.39 (3.489) | 24.12 (3.786) | 23.57 (3.578)

OUTCOME MEASURES:

1. Primary Outcome: Rabies Virus Neutralizing Activity (RVNA) of Geometric Mean Concentration (GMC) at Study Day 8
Description: Rabies Virus Neutralizing Activity (RVNA) was assessed using Rapid Fluorescent Focus Inhibition Test (RFFIT).
Time Frame: Day 8
Population: The primary analysis set of the outcome measure data is Per-Protocol Analysis Set (PPS). The PPS included all subjects who were randomized, received the correct study drug, passed the confirmation of the inclusion/exclusion criteria *, completed the rabies vaccination schedule as required by the protocol on Day 29 of the study, had no major protocol violations impacting efficacy evaluation, received adequate wound treatment of all exposed sites, and received study drug injection.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Experimental Group: SYN023+Rabies Vaccine | Control Group: Human Rabies Immune Globulin (HRIG)+Rabie Vaccine
Number analyzed (Participants) | 507 | 165
IU/mL | 4.346 [4.111 to 4.595] | 0.232 [0.198 to 0.271]

2. Primary Outcome: Number of Probable or Confirmed Rabies Cases
Description: WHO's Classification of Rabies Cases:
  1. Suspected case: refers to a case that satisfies the definition of clinical case;
  2. Probable case: refers to a suspected case with a reliable medical history of contact with any suspected animal infected with the rabies virus;
  3. Confirmed case: refers to a suspected or probable case that is proved to be infected based on the lab test result.
Time Frame: Day 1 to Day 365
Measure: Number; unit: participants
Arm/Group | Experimental Group: SYN023+Rabies Vaccine | Control Group: Human Rabies Immune Globulin (HRIG)+Rabie Vaccine
Number analyzed (Participants) | 750 | 250
participants | 0 | 0

3. Secondary Outcome: Rabies Virus Neutralizing Activity (RVNA) of Geometric Mean Concentration (GMC)
Description: Rabies Virus Neutralizing Activity (RVNA) was assessed using Rapid Fluorescent Focus Inhibition Test (RFFIT).
Time Frame: Days 4, 15, 43, 99, 183 and 365
Population: The analysis set of the outcome measure data is Per-Protocol Analysis Set (PPS). The PPS included all subjects who were randomized, received the correct study drug, passed the confirmation of the inclusion/exclusion criteria *, completed the rabies vaccination schedule as required by the protocol on Day 29 of the study, had no major protocol violations impacting efficacy evaluation, received adequate wound treatment of all exposed sites, and received study drug injection.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Experimental Group: SYN023+Rabies Vaccine | Control Group: Human Rabies Immune Globulin (HRIG)+Rabie Vaccine
Number analyzed (Participants) | 507 | 165
IU/mL
  Day 4 | 4.212 [3.962 to 4.479] | 0.193 [0.172 to 0.216]
  Day 15 | 13.590 [12.624 to 14.630] | 7.651 [6.241 to 9.380]
  Day 43: number analyzed (Participants) | 503 | 165
  Day 43 | 13.084 [12.238 to 13.989] | 16.003 [13.650 to 18.762]
  Day 99: number analyzed (Participants) | 495 | 161
  Day 99 | 2.023 [1.869 to 2.190] | 5.108 [4.109 to 6.351]
  Day 183: number analyzed (Participants) | 496 | 160
  Day 183 | 0.891 [0.812 to 0.978] | 3.319 [2.681 to 4.108]
  Day 365: number analyzed (Participants) | 483 | 160
  Day 365 | 0.520 [0.473 to 0.572] | 1.645 [1.343 to 2.014]

4. Secondary Outcome: Percentage of Participants With Rabies Virus Neutralizing Activity (RVNA) ≥0.5 IU/mL
Description: Rabies Virus Neutralizing Activity (RVNA) was assessed using Rapid Fluorescent Focus Inhibition Test (RFFIT).
Time Frame: Days 4, 8, 15, 43, 99, 183 and 365
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants(%)
Arm/Group | Experimental Group: SYN023+Rabies Vaccine | Control Group: Human Rabies Immune Globulin (HRIG)+Rabie Vaccine
Number analyzed (Participants) | 507 | 165
percentage of participants(%)
  Day 4 | 99.8 [98.906 to 99.995] | 9.1 [5.178 to 14.551]
  Day 8 | 99.6 [98.582 to 99.952] | 17.6 [12.098 to 24.256]
  Day 15 | 100 [99.275 to 100] | 96.4 [92.253 to 98.654]
  Day 43: number analyzed (Participants) | 503 | 165
  Day 43 | 100 [98.269 to 100] | 99.4 [96.670 to 99.985]
  Day 99: number analyzed (Participants) | 495 | 161
  Day 99 | 97.8 [96.059 to 98.886] | 97.5 [93.761 to 99.319]
  Day 183: number analyzed (Participants) | 496 | 160
  Day 183 | 72.8 [68.636 to 76.654] | 95.6 [91.194 to 98.223]
  Day 365: number analyzed (Participants) | 483 | 160
  Day 365 | 47.2 [42.678 to 51.766] | 81.9 [75.018 to 87.513]

5. Secondary Outcome: Area Under the Efficacy Curve for the Geometric Mean Concentration (GMC) of Rabies Virus Neutralizing Activity (RVNA)
Description: Rabies Virus Neutralizing Activity (RVNA) was assessed using Rapid Fluorescent Focus Inhibition Test (RFFIT). Area Under the Efficacy Curve for the GMC of RVNA from Study Day 1 to Day 15 after administration (AUEC1-15)
Time Frame: Day 1 to Day 15
Population: The Per Protocol Set (PPS) included all subjects who were randomized, received the correct study drug, passed the confirmation of the inclusion/exclusion criteria *, completed the rabies vaccination schedule as required by the protocol on Day 29 of the study, had no major protocol violations impacting efficacy evaluation, received adequate wound treatment of all exposed sites, and received study drug injection.
Measure: Geometric Mean (95% Confidence Interval); unit: days *IU/mL
Arm/Group | Experimental Group: SYN023+Rabies Vaccine | Control Group: Human Rabies Immune Globulin (HRIG)+Rabie Vaccine
Number analyzed (Participants) | 507 | 165
days *IU/mL | 96.972 [91.955 to 102.263] | 31.869 [26.563 to 38.233]

ADVERSE EVENTS:
Time Frame: 365 days
Groups:
- Experimental Group: SYN023+Rabies Vaccine: 1000 patients aged 18 and above with WHO Category III rabies exposure should be enrolled as planned and randomly assigned to the experimental group and the control group based on a ratio of 3:1 through on-site stratification as part of PEP.
  SYN023: 0.3 mg/kg, wound infiltration injection. If the study drug isn't used up after infiltration injection for all wounds, the remaining amount should be injected into the muscles far away from the vaccine injection sites Frequency/duration: at Day 1
  Rabies Vaccine: 0.5 mL, intramuscular injection into the deltoid muscle Frequency/duration: at Day 1, 4, 8, 15, 29
- Control Group: HRIG+Rabie Vaccine: 1000 patients aged 18 and above with WHO Category III rabies exposure should be enrolled as planned and randomly assigned to the experimental group and the control group based on a ratio of 3:1 through on-site stratification as part of PEP.
  HRIG: 20 IU/kg, wound infiltration injection. If the study drug isn't used up after infiltration injection for all wounds, the remaining amount should be injected into the muscles far away from the vaccine injection sites Frequency/duration: at Day 1
  Rabies Vaccine: 0.5 mL, intramuscular injection into the deltoid muscle Frequency/duration: at Day 1, 4, 8, 15, 29
Arm/Group | Experimental Group: SYN023+Rabies Vaccine | Control Group: HRIG+Rabie Vaccine
All-Cause Mortality (participants affected / at risk) | 0/750 | 0/250
Serious Adverse Events (participants affected / at risk) | 41/750 | 14/250
Other Adverse Events (participants affected / at risk) | 315/750 | 138/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Group: SYN023+Rabies Vaccine (N=750) | Control Group: HRIG+Rabie Vaccine (N=250)
Infectious pneumonitis (Infections and infestations) | 4 (4) | 2 (2)
Herpes zoster (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Bacterial pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0)
Scrub typhus (Infections and infestations) | 0 (0) | 1 (2)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Urethritis (Infections and infestations) | 1 (1) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0)
Ureteritis (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Infected bite (Infections and infestations) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 2 (3) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hypertrophic anal papilla (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusions (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral Trauma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Brain herniation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Snake bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cerebral hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral hypoperfusion (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Ischial neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Vertebral end plate inflammation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ureteral calculus (Renal and urinary disorders) | 4 (4) | 0 (0)
Renal hydrocele (Renal and urinary disorders) | 3 (3) | 0 (0)
Nephrolith (Renal and urinary disorders) | 3 (3) | 0 (0)
Renal Colic (Renal and urinary disorders) | 2 (2) | 0 (0)
Hydroureter (Renal and urinary disorders) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough variant asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Neonatal aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neonatal hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma lung stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carcinoid tumour of the gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia newborn (Hepatobiliary disorders) | 1 (1) | 0 (0)
Shoulder dystocia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
hypersensitivity reaction (Immune system disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Allergic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Aortic valve disease mixed (Cardiac disorders) | 1 (1) | 0 (0)
Vein varicose (Vascular disorders) | 0 (0) | 1 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Group: SYN023+Rabies Vaccine (N=750) | Control Group: HRIG+Rabie Vaccine (N=250)
Administration site swelling (General disorders) | 128 | 87
Administration site pain (General disorders) | 36 | 20
Administration site erythema (General disorders) | 32 | 15
Administration site pruritus (General disorders) | 7 | 6
Administration site haemorrhage (General disorders) | 6 | 0
Administration site paraesthesia (General disorders) | 1 | 1
Vaccination site pain (General disorders) | 27 | 12
Vaccination site Pruritus (General disorders) | 2 | 3
Vaccination site discomfort (General disorders) | 1 | 0
Vaccination site rash (General disorders) | 0 | 1
Vaccination site swelling (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 1 | 0
Fever (General disorders) | 17 | 7
Asthenia (General disorders) | 4 | 3
Chills (General disorders) | 3 | 2
Chest pain (General disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 6
Running nose (Respiratory, thoracic and mediastinal disorders) | 9 | 5
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 3
nasal congestion. (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Headache (Nervous system disorders) | 30 | 12
Dizziness (Nervous system disorders) | 12 | 4
Hypaesthesia (Nervous system disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 11 | 6
Nasopharyngitis (Infections and infestations) | 9 | 1
Infected bite (Infections and infestations) | 2 | 1
Gastroenteritis (Infections and infestations) | 2 | 0
Pericoronitis (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 5 | 4
Nausea (Gastrointestinal disorders) | 3 | 3
Toothache (Gastrointestinal disorders) | 5 | 1
Hemorrhoids (Gastrointestinal disorders) | 2 | 1
Mouth ulceration (Gastrointestinal disorders) | 2 | 3
Bloating (Gastrointestinal disorders) | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Epigastric pain (Gastrointestinal disorders) | 1 | 2
Noninfective gingivitis (Gastrointestinal disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0
Dental caries (Gastrointestinal disorders) | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Dental paraesthesia (Gastrointestinal disorders) | 0 | 1
Gingival swelling (Gastrointestinal disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 2
Limb pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Vertebral wedging (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone hypertrophy (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 3 | 1
Animal scratches (Injury, poisoning and procedural complications) | 1 | 1
Skin injury (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous hematoma (Injury, poisoning and procedural complications) | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Inflammation of wound (Injury, poisoning and procedural complications) | 1 | 0
Injection related reaction (Injury, poisoning and procedural complications) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 2
Rash (Skin and subcutaneous tissue disorders) | 5 | 0
Allergic dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Urticarial rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 6 | 2
Pallor (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 1 | 0
Aortic dilatation (Vascular disorders) | 1 | 0
Nephrolith (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 1
Urgency urination (Renal and urinary disorders) | 1 | 0
Frequent Micturition (Renal and urinary disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Blood pressure increased (Investigations) | 2 | 0
Spinal X-ray abnormal (Investigations) | 1 | 0
Ultrasound prostate abnormal (Investigations) | 1 | 0
Blood zinc abnormal (Investigations) | 0 | 1
Breast hyperplasia (Reproductive system and breast disorders) | 2 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0
Hypomenorrhoea (Reproductive system and breast disorders) | 1 | 0
Gallbladder polyp (Hepatobiliary disorders) | 2 | 0
Fatty degeneration of liver (Hepatobiliary disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Atrial enlargement (Cardiac disorders) | 1 | 0
Palpitation (Cardiac disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Poor quality sleep (Psychiatric disorders) | 1 | 0
Fear of injection (Psychiatric disorders) | 1 | 0
Dry eyes (Eye disorders) | 0 | 1
Hyperaemia of conjunctiva (Eye disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Tracheal operation (Surgical and medical procedures) | 1 | 0
Accessory breast (Congenital, familial and genetic disorders) | 1 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT04644484/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-04): https://cdn.clinicaltrials.gov/large-docs/84/NCT04644484/SAP_001.pdf